CLINICAL TRIAL: NCT06216639
Title: EU4Health Project Eurohelican: A Single-center Prospective Feasibility Study of the Proposed Test-and-treat Preventive Screening Program in Younger Slovenian Participants Aged 30-34 Years With or Without Helicobacter Pylori Infection
Brief Title: Feasibility Study of the Proposed Test-and-treat Screening Program in Younger Participants With H. Pylori Infection
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Public Health, Slovenia (Other Government)
Collaborators: Community Healthcare Center dr. Adolf Drolc Maribor (HCM) (Other)
Responsible Party: Sponsor
Other Study IDs: EUROHELICAN01
Record Dates: First submitted 2024-01-05; First posted 2024-01-22 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; Stomach Neoplasms; Mass Screening; Preventive Health Services; Feasibility Studies; Screening Acceptability; Treatment Outcome; Test-and-treat Strategy; Drug-Related Side Effects and Adverse Reactions
MeSH Terms: conditions — Stomach Neoplasms; Drug-Related Side Effects and Adverse Reactions | interventions — bismuth tripotassium dicitrate; Esomeprazole; Metronidazole; Amoxicillin; Clarithromycin; Levofloxacin; Ofloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals between 30 and 34 years of age registered at HCM: Random sample of participants representing the eligible cohort is drawn.
  Interventions: Drug: Bismuth Subcitrate; Drug: Esomeprazole; Drug: Metronidazole; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Levofloxacin

INTERVENTIONS:
Drug: Bismuth Subcitrate — Tripotassium dicitratobismuthate 120 mg film-coated tablets. Prescribed for both primary and (potential) secondary treatment with bismuth-based quadruple therapy in participants with active H. pylori infection. The prescribed daily dose is 120 mg QID for a period of 14 days.
  Other Names: Bizmutov oksid Krka 120 mg filmsko obložene tablete
Drug: Esomeprazole — Esomeprazol 40 mg gastro-resistant tablets or hard capsules. Which one of the three brands is prescribed for an individual participant in this prospective study depends on the decision of a chosen personal physician. Prescribed for both primary and (potential) secondary treatment with bismuth-based quadruple therapy in participants with active H. pylori infection. The prescribed daily dose is 40 mg BID for a period of 14 days.
  Other Names: Emozul 40 mg trde gastrorezistentne kapsule; Nexium 40 mg gastrorezistentne tablete; Nillar 40 mg gastrorezistentne tablete
Drug: Metronidazole — Metronidazol 400 mg tablets. Prescribed for both primary and (potential) secondary treatment with bismuth-based quadruple therapy in participants with active H. pylori infection. The prescribed daily dose is 400 mg QID for a period of 14 days.
  Other Names: Efloran 400 mg tablete
Drug: Amoxicillin — Amoxicillin 500 mg dispersible tablets or hard capsules. Which one of the two brands is prescribed for an individual participant in this prospective study depends on the decision of a chosen personal physician. Prescribed only for the primary treatment with bismuth-based quadruple therapy in participants with active H. pylori infection who are not allergic to penicillin. The prescribed daily dose is 500 mg QID for a period of 14 days.
  Other Names: Amoksicilin Belupo 500 mg disperzibilne tablete; Hiconcil 500 mg trde kapsule
Drug: Clarithromycin — Clarithromycin 500 mg film-coated tablets. Prescribed only for the primary treatment with bismuth-based quadruple therapy in participants with active H. pylori infection who are allergic to penicillin. The prescribed daily dose is 500 mg BID for a period of 14 days.
  Other Names: Fromilid 500 mg filmsko obložene tablete
Drug: Levofloxacin — Levofloxacin 500 mg film-coated tablets. Prescribed only for the (potential) secondary treatment with bismuth-based quadruple therapy in participants with active H. pylori infection. The prescribed daily dose is 500 mg OID for a period of 14 days.
  Other Names: Tavanic 500 mg filmsko obložene tablete

SUMMARY:
This prospective non-interventional study is being conducted as part of the EU4Health project Eurohelican. The main goal of this pilot study is to evaluate the feasibility and acceptability of implementing the proposed "test-and-treat" screening program on a population-based sample. Participants will be randomly selected from a younger population registered at the primary level of care and tested for the presence of active infection with Helicobacter pylori (H. pylori). Infected participants will undergo a bismuth-based quadruple treatment with antibiotics and a proton pump inhibitor, and will be controlled for eradication success by taking the urea breath test (UBT). A number of other participant outcomes will be also measured to provide additional pro et contra argumentation for the potential future implementation of a population-based test-and-treat screening program in Slovenia. Research reports will be disseminated and results will be presented to the public and scientific community to foster future developments in gastric cancer prevention.

DETAILED DESCRIPTION:
Gastric cancer remains an important public health issue due to its high incidence rate and relatively low five-year survival rate. H. pylori infection has been found to be the main cause of gastric cancer and is responsible for 89% of non-cardia gastric cancers. There is also evidence that H. pylori eradication significantly reduces the incidence and mortality due to gastric cancer. According to the proposal based on available data, the population-based test-and-treat screening program may be the best available evidence-based intervention to prevent the occurrence of gastric cancer. In its recommendations from September 9th 2023, the European Council also supported the implementation of a screening program particularly in European regions with an increased prevalence of H. pylori and incidence of gastric cancer. The aim of this study is to scientifically evaluate the feasibility, acceptability and effectiveness of the proposed population-based test-and-treat strategy for the eradication of H. pylori infection.

The proposed test-and-treat strategy is targeted at the population around the age of 30 years who are infected with H. pylori and predominantly asymptomatic. The main questions it aims to answer are:

* Is the proposed population-based H. pylori test-and-treat strategy feasible and acceptable in a community health service setting?
* Is the proposed population-based H. pylori test-and-treat strategy effective in a community health service setting?
* What is the profile of adverse events in the treated participants?

Participants will be randomly selected from the population pool of individuals aged 30-34 years who have a chosen personal physician at Community Healthcare Center dr. Adolf Drolc Maribor (HCM). Enrolled participants who will give their informed consent will be interviewed by a registered nurse regarding risk factors for developing H. pylori infection and selected lifestyle habits. In addition, serology testing for the presence of H. pylori antibodies will be performed on all participants. Participants with a positive serology result will be given a confirmatory urea breath test (UBT). Those participants with a confirmed active H. pylori infection will be treated with bismuth-based quadruple therapy, and the success of eradication will then be verified by UBT one month after the treatment. Participants with a positive result of the second UBT will be treated again with a second-line modified bismuth-based quadruple therapy, and the success of eradication will be verified by UBT. Compliance with testing and treatment, treatment outcomes, adverse events and reasons for withdrawing participation will be monitored for each of the participants. The feasibility and sustainability of the proposed test-and-treat strategy will be evaluated using several key performance indicators that follow the structure of five principal areas of feasibility. Data will be entered into the REDCap online survey application and analyzed using IBM SPSS Statistics software.

The results of this study will enable to potentially scale up the project to the national level and present a potential model for the implementation of this strategy in Europe. Second, the results will contribute to the implementation of the Europe's Beating Cancer Plan goal of preventing gastric cancers caused by H. pylori infections. Finally, this study will provide additional real-world data for the preparation of Expert Working Group Report of the International Agency for Research on Cancer of the World Health Organization (IARC/WHO), which will include a minimum set of standards for the implementation of a population-based screening program at the international level.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 30-34 years,
* Individuals who have a chosen personal physician at HCM,
* Individuals who sign an informed consent to participate, and
* Individuals who do not have a congenital or acquired intellectual disability.

Exclusion Criteria:

* Individuals younger than 30 years or older than 34 years,
* Individuals who do not have a chosen personal physician at HCM,
* Individuals who do not sign informed consent for participation,
* Individuals with intellectual or developmental limitations who are unable to provide a fully-informed consent to participate (based on the assessment of the patient's primary care team)
* Individuals who were previously treated for H. pylori infection, and
* Individuals with a history of partial of total gastric resection due to benign or malign lesions.

Ages: 30 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The primary pool of potential participants is composed of younger individuals of both sexes between 30 and 34 years of age with a registered chosen personal physician at HCM. A single non-interventional cohort of 4,000 individuals will be randomly selected using Monte-Carlo sampling method. All selected individuals in a sample will be invited to participate. If the individual expresses interest in participating, the primary care team staff will decide whether or not to enroll the individual in the study based on the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Healthcare workers' assessment of feasibility and acceptability of the proposed practical implementation of a screening program | 1 year after the completion of prospective study.
  Responses to qualitative questions and summary statistics from a post-enrollment questionnaire for healthcare workers involved into the implementation of the screening program. The questionnaires will be completed by up to 100 chosen personal physicians and registered nurses from HCM who participated in this prospective study. Questionnaire preparation follows the key performance indicators for assessing the five dimensions of the standardized TELOS framework of project feasibility.

SECONDARY OUTCOMES:
Participation rate of subjects selected for the program | 3 months after: a) completion of the enrollment process (points a)-d)); b) completion of the prospective study (points e)-h)).
  Subtraction of 1) study participants who:
  1. did not respond to an invitation,
  2. signed the informed consent form but were not included in the study due to exclusion criteria,
  3. declined to take a serology test,
  4. declined to take any of the UBTs as specified in the study protocol,
  5. had their therapy postponed due to maternity reasons,
  6. declined to be re-treated after the treatment failure of primary therapy,
  7. voluntarily withdrew at any time during their participation in the study,
  8. withdrew from the study within points a)-g) combined,
  from 2) all participants invited in the study.
  The participation rate is measured in frequencies and percentage points (%).
Eradication rate of infection with H. pylori | 3 months after enrollment of the last participant who took a control UBT after the completion of primary bismuth-based quadruple therapy regimen.
  Subtraction of 1) participants who were subjected to treatment failure of the primary therapy regimen from 2) all participants with an active H. pylori infection who underwent the primary bismuth-based quadruple therapy regimen.
  The eradication rate is measured in frequencies and percentage points (%).
Description of the adverse events profile | 6 months after enrollment of the last participant who took a second control UBT after the completion of secondary bismuth-based quadruple therapy regimen.
  Qualitative records of all self-reported (or physician-reported) adverse events during and after primary (or secondary) bismuth-based quadruple therapy regimen. All non-serious or serious adverse event will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Tepeš, PhD, Study Director — NIJZ; Jernej Završnik, PhD, Principal Investigator — Community Healthcare Center dr. Adolf Drolc Maribor (HCM)
Locations (1):
- Community Healthcare Center dr. Adolf Drolc Maribor (HCM), Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Chiang TH, Chang WJ, Chen SL, Yen AM, Fann JC, Chiu SY, Chen YR, Chuang SL, Shieh CF, Liu CY, Chiu HM, Chiang H, Shun CT, Lin MW, Wu MS, Lin JT, Chan CC, Graham DY, Chen HH, Lee YC. Mass eradication of Helicobacter pylori to reduce gastric cancer incidence and mortality: a long-term cohort study on Matsu Islands. Gut. 2021 Feb;70(2):243-250. doi: 10.1136/gutjnl-2020-322200. Epub 2020 Aug 13. PMID 32792335
- [Background] de Martel C, Georges D, Bray F, Ferlay J, Clifford GM. Global burden of cancer attributable to infections in 2018: a worldwide incidence analysis. Lancet Glob Health. 2020 Feb;8(2):e180-e190. doi: 10.1016/S2214-109X(19)30488-7. Epub 2019 Dec 17. PMID 31862245
- [Background] Ford AC, Yuan Y, Moayyedi P. Helicobacter pylori eradication therapy to prevent gastric cancer: systematic review and meta-analysis. Gut. 2020 Dec;69(12):2113-2121. doi: 10.1136/gutjnl-2020-320839. Epub 2020 Mar 23. PMID 32205420
- [Background] Kowada A. A Population-Based Helicobacter pylori Eradication Strategy Is More Cost-Effective than Endoscopic Screening. Dig Dis Sci. 2023 May;68(5):1735-1746. doi: 10.1007/s10620-022-07795-z. Epub 2022 Dec 24. PMID 36565366
- [Background] Lansdorp-Vogelaar I, Sharp L. Cost-effectiveness of screening and treating Helicobacter pylori for gastric cancer prevention. Best Pract Res Clin Gastroenterol. 2013 Dec;27(6):933-47. doi: 10.1016/j.bpg.2013.09.005. Epub 2013 Sep 27. PMID 24182612
- [Background] Lee YC, Chiang TH, Liou JM, Chen HH, Wu MS, Graham DY. Mass Eradication of Helicobacter pylorito Prevent Gastric Cancer: Theoretical and Practical Considerations. Gut Liver. 2016 Jan;10(1):12-26. doi: 10.5009/gnl15091. PMID 26696028
- [Background] Lee YC, Chiang TH, Chou CK, Tu YK, Liao WC, Wu MS, Graham DY. Association Between Helicobacter pylori Eradication and Gastric Cancer Incidence: A Systematic Review and Meta-analysis. Gastroenterology. 2016 May;150(5):1113-1124.e5. doi: 10.1053/j.gastro.2016.01.028. Epub 2016 Feb 2. PMID 26836587
- [Background] Liou JM, Malfertheiner P, Lee YC, Sheu BS, Sugano K, Cheng HC, Yeoh KG, Hsu PI, Goh KL, Mahachai V, Gotoda T, Chang WL, Chen MJ, Chiang TH, Chen CC, Wu CY, Leow AH, Wu JY, Wu DC, Hong TC, Lu H, Yamaoka Y, Megraud F, Chan FKL, Sung JJ, Lin JT, Graham DY, Wu MS, El-Omar EM; Asian Pacific Alliance on Helicobacter and Microbiota (APAHAM). Screening and eradication of Helicobacter pylori for gastric cancer prevention: the Taipei global consensus. Gut. 2020 Dec;69(12):2093-2112. doi: 10.1136/gutjnl-2020-322368. Epub 2020 Oct 1. PMID 33004546
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Background] Malfertheiner P, Megraud F, Rokkas T, Gisbert JP, Liou JM, Schulz C, Gasbarrini A, Hunt RH, Leja M, O'Morain C, Rugge M, Suerbaum S, Tilg H, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study group. Management of Helicobacter pylori infection: the Maastricht VI/Florence consensus report. Gut. 2022 Aug 8:gutjnl-2022-327745. doi: 10.1136/gutjnl-2022-327745. Online ahead of print. PMID 35944925
- [Background] Ozeki K, Asano M, Furuta T, Ojima T. Relationship between primary eradication of Helicobacter pylori and drinking habits in women: collaborative research between a pharmacy and a clinic. Epidemiol Infect. 2019 Oct 22;147:e292. doi: 10.1017/S0950268819001730. PMID 31637982
- [Background] Park JY, Herrero R. Recent progress in gastric cancer prevention. Best Pract Res Clin Gastroenterol. 2021 Mar-Apr;50-51:101733. doi: 10.1016/j.bpg.2021.101733. Epub 2021 Feb 18. PMID 33975687
- [Background] Sarmasti M, Khoshbaten M, Khalili F, Yousefi M. Cost-Effectiveness of Screening Helicobacter pylori for Gastric Cancer Prevention: a Systematic Review. J Gastrointest Cancer. 2022 Dec;53(4):1093-1103. doi: 10.1007/s12029-021-00726-7. Epub 2021 Oct 25. PMID 34694594
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Tan Y, Wei Z, Liu K, Qin Y, Hui W. Lifestyle habits and gastric cancer in an East Asian population: a Mendelian randomization study. Front Oncol. 2023 Sep 4;13:1224753. doi: 10.3389/fonc.2023.1224753. eCollection 2023. PMID 37731647
- [Background] Yu J, Yang P, Qin X, Li C, Lv Y, Wang X. Impact of smoking on the eradication of Helicobacter pylori. Helicobacter. 2022 Feb;27(1):e12860. doi: 10.1111/hel.12860. Epub 2021 Oct 27. PMID 34708484